CLINICAL TRIAL: NCT04733547
Title: Spectral Analysis of Central Venous Pressure Waveform in Patients Undergoing Donor Hepatectomy
Brief Title: Spectral Analysis of Central Venous Pressure Waveform
Status: Completed | Type: Observational
Sponsor: JongHae Kim (Other)
Responsible Party: Sponsor-Investigator, JongHae Kim, Professor, Daegu Catholic University Medical Center
Organization: Daegu Catholic University Medical Center (Other)
Other Study IDs: CR-21-007
Record Dates: First submitted 2021-01-26; First posted 2021-02-02 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Donor Hepatectomy; Central Venous Catheter; Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Donor hepatectomy: Live donors undergoing hepatectomy
  Interventions: Procedure: Placement of a central venous catheter; Device: Monitoring of central venous pressure; Drug: Furosemide-induced hypovolemia before graft procurement; Drug: Replacement of fluid loss after graft procurement; Device: Monitoring of stroke volume variation

INTERVENTIONS:
Procedure: Placement of a central venous catheter — The right internal jugular vein is located at the first rib level under ultrasound-guidance. Using an out-of-plane technique, a needle is introduced into the lumen of the vessel. The aspiration of blood into the syringe connected to the hub of the needle confirms the placement of the needle tip in the lumen. After the syringe is detached from the needle, a guidewire is advanced into the vessel lumen through the needle. A dilator is introduced over the guidewire and subsequently is removed. Then, a central venous catheter is introduced over the guidewire into the vessel lumen through the pathway expanded by the dilator. The catheter tip is placed in the superior vena cava by inserting the catheter as far as the distance between the edge of the right transverse process of the first thoracic vertebra and the carina, which is preoperatively measured on a posteroanterior chest radiograph.
Device: Monitoring of central venous pressure — Following the placement of a central venous catheter, a fluid-filled system for monitoring central venous pressure is connected to the proximal lumen of the catheter. The reference transducer is placed at the level of 4/5 of the anteroposterior diameter of the thorax.
Drug: Furosemide-induced hypovolemia before graft procurement — Patients fast from 10 pm the day before surgery. On the arrival at the operating room, an intravenous catheter for Plasmalyte infusion is placed into the right cephalic or basilic vein. The distal lumen of the central venous catheter is used for the infusion of 6% hydroxyethyl starch. Fluid requirements due to anesthesia, surgery, and no per os intake are not replaced by minimizing the administration of the fluids. Five minutes after the collection of the baseline data, 20 mg of furosemide is administered to promote diuresis for facilitating the venous outflow of the liver. An additional dose of furosemide 20 mg is given if the urine output is <1 ml/kg within 30 minutes after the first dose. Unless the second dose of furosemide produces >1 ml/kg of urine within 30 minutes, 40 mg of furosemide is administered. In the absence of effective diuresis (1 ml/kg within 30 minutes after each dose), the use of furosemide is abandoned and the patients are excluded from the study.
Drug: Replacement of fluid loss after graft procurement — Immediately after the graft procurement, 500 ml of 6% hydroxyethyl starch are infused over 25 minutes. Afterward, Plasmalyte is infused at a rate of 10 ml/min until the end of surgery.
Device: Monitoring of stroke volume variation — Following anesthesia induction, the right radial artery is catheterized. The catheter is connected to the EV1000 monitor (Edwards Lifesciences, Irvine, CA) through the FloTrac transducer (Edwards Lifesciences). The transducer is level with the one for central venous pressure monitoring. Using pulse contour analysis without external calibration, the stroke volume for each heartbeat is measured. At a 20-second interval, stroke volume variation is calculated as (maximum stroke volume - minimum stroke volume)/mean stroke volume.

SUMMARY:
The use of central venous pressure has been abandoned for the assessment of intravascular volume status. The dynamic fluctuation of central venous pressure according to heart rate is quantitatively measured by spectral analysis of the central venous pressure waveform. Its clinical utility in the assessment of intravascular volume status is investigated.

DETAILED DESCRIPTION:
The use of central venous pressure, which is one of the static preload indices, has been abandoned for the assessment of intravascular volume status because of its unreliability. The static preload indices have been replaced with dynamic preload indices, such as stroke volume variation or pulse pressure variation because the dynamic preload indices reliably predict fluid responsiveness and perform better than the static preload indices. However, the periodic component of central venous pressure, which goes with cardiac cycles, has not been investigated. The power corresponding to heart rate from spectral analysis of central venous pressure waveform represents the extent of the dynamic fluctuation of central venous pressure and is assumed to reflect intravascular volume status. It is hypothesized that the spectral power of central venous pressure corresponding to heart rate represents intravascular volume status.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1
* Scheduled for donor hepatectomy under general anesthesia

Exclusion Criteria:

* Arrhythmia
* Valvular heart disease
* Coronary artery disease
* Cerebrovascular disease
* Hypertension
* Diabetes mellitus
* Renal insufficiency
* Pulmonary problems
* Any type of liver disease
* Body mass index greater than 35 kg/m2
* Human immunodeficiency virus infection
* Psychosocial problems
* Electrolyte imbalance
* Reoperation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients are recruited from a tertiary university hospital
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Spectral power of central venous pressure corresponding to heart rate during 5 minutes before graft procurement | During 5 minutes before graft procurement
  A band-pass filter (0.15-3 Hz) is applied to the 5 minute-long segment. The 5 minute-long segments are divided into 100 second-long segments overlapping 50% with each adjacent segment. Each segment is submitted to fast Fourier transformation. The spectral powers obtained from the periodograms of each segment are averaged. The integrated area corresponding to heart rate is the spectral power corresponding to heart rate.

SECONDARY OUTCOMES:
Spectral powers of central venous pressure corresponding to respiratory rate and heart rate during 5 minutes before the first dose of furosemide | During 5 minutes before the first dose of furosemide
  A band-pass filter (0.15-3 Hz) is applied to the 5 minute-long segment. The 5 minute-long segments are divided into 100 second-long segments overlapping 50% with each adjacent segment. Each segment is submitted to fast Fourier transformation. The spectral powers obtained from the periodograms of each segment are averaged. The integrated areas corresponding to respiratory rate and heart rate are the spectral powers corresponding to respiratory rate and heart rate.
Spectral powers of central venous pressure corresponding to respiratory rate and heart rate between 30 and 35 minutes after surgical incision | Between 30 and 35 minutes after surgical incision
  A band-pass filter (0.15-3 Hz) is applied to the 5 minute-long segment. The 5 minute-long segments are divided into 100 second-long segments overlapping 50% with each adjacent segment. Each segment is submitted to fast Fourier transformation. The spectral powers obtained from the periodograms of each segment are averaged. The integrated areas corresponding to respiratory rate and heart rate are the spectral powers corresponding to respiratory rate and heart rate.
Spectral power of central venous pressure corresponding to respiratory rate during 5 minutes before graft procurement | During 5 minutes before graft procurement
  A band-pass filter (0.15-3 Hz) is applied to the 5 minute-long segment. The 5 minute-long segments are divided into 100 second-long segments overlapping 50% with each adjacent segment. Each segment is submitted to fast Fourier transformation. The spectral powers obtained from the periodograms of each segment are averaged. The integrated area corresponding to respiratory rate is the spectral power corresponding to respiratory rate.
Spectral powers of central venous pressure corresponding to respiratory rate and heart rate during 5 minutes after administration of 6% hydroxyethyl starch | During 5 minutes after administration of 6% hydroxyethyl starch
  A band-pass filter (0.15-3 Hz) is applied to the 5 minute-long segment. The 5 minute-long segments are divided into 100 second-long segments overlapping 50% with each adjacent segment. Each segment is submitted to fast Fourier transformation. The spectral powers obtained from the periodograms of each segment are averaged. The integrated areas corresponding to respiratory rate and heart rate are the spectral powers corresponding to respiratory rate and heart rate.
Stroke volume variation during 5 minutes before the first dose of furosemide | During 5 minutes before the first dose of furosemide
  The median of the values calculated at a 20-second interval
Stroke volume index during 5 minutes before the first dose of furosemide | During 5 minutes before the first dose of furosemide
  The median of the values calculated at a 20-second interval
Cardiac index during 5 minutes before the first dose of furosemide | During 5 minutes before the first dose of furosemide
  The median of the values calculated at a 20-second interval
Stroke volume variation between 30 and 35 minutes after surgical incision | Between 30 and 35 minutes after surgical incision
  The median of the values calculated at a 20-second interval
Stroke volume index between 30 and 35 minutes after surgical incision | Between 30 and 35 minutes after surgical incision
  The median of the values calculated at a 20-second interval
Cardiac index between 30 and 35 minutes after surgical incision | Between 30 and 35 minutes after surgical incision
  The median of the values calculated at a 20-second interval
Stroke volume variation during 5 minutes before graft procurement | During 5 minutes before graft procurement
  The median of the values calculated at a 20-second interval
Stroke volume index during 5 minutes before graft procurement | During 5 minutes before graft procurement
  The median of the values calculated at a 20-second interval
Cardiac index during 5 minutes before graft procurement | During 5 minutes before graft procurement
  The median of the values calculated at a 20-second interval
Stroke volume variation during 5 minutes after administration of 6% hydroxyethyl starch | During 5 minutes after administration of 6% hydroxyethyl starch
  The median of the values calculated at a 20-second interval
Stroke volume index during 5 minutes after administration of 6% hydroxyethyl starch | During 5 minutes after administration of 6% hydroxyethyl starch
  The median of the values calculated at a 20-second interval
Cardiac index during 5 minutes after administration of 6% hydroxyethyl starch | During 5 minutes after administration of 6% hydroxyethyl starch
  The median of the values calculated at a 20-second interval
Total dose of furosemide | At graft procurement
  The total dose of furosemide used for the promotion of diuresis
Urine output at graft procurement | At graft procurement
  The total amount of urine output between the placement of urinary catheter and graft procurement
Total urine output at the end of surgery | At the end of surgery
  The total amount of urine output at the end of surgery
Intraoperative blood loss | 1 day after surgery
  Calculated as blood loss (ml) = [estimated blood volume*(preoperative hematocrit-postoperative hematocrit)]/mean between the 2 hematocrit values, where estimated blood volume (ml) = weight(kg)^0.425*height(cm)^0.725*0.007184*2217+age(years)*1.06 for female and weight(kg)^0.425*height(cm)^0.725*0.007184*3064-825 for male

OTHER OUTCOMES:
Age | On arrival at the operating room
  Age at the time of surgery
Sex | On arrival at the operating room
  Biological sex
Height | The day before surgery
  Measured in cm
Weight | The day before surgery
  Measured in kg
Aspartate transaminase | The day before surgery
  Measured in U/L
Alanine transaminase | The day before surgery
  Measured in U/L
Blood urea nitrogen | The day before surgery
  Measured in mg/dl
Creatinine | The day before surgery
  Measured in mg/dl
Serum sodium level | The day before surgery
  Measured in mmol/L
Serum potassium level | The day before surgery
  Measured in mmol/L
Serum chloride level | The day before surgery
  Measured in mmol/L
Graft weight | At graft procurement
  Measured in gram
Total amount of fluids | At the end of surgery
  The total volume of colloids and crystalloids administered throughout the entire surgery
Aspartate transaminase | 1 hour after surgery
  Measured in U/L
Alanine transaminase | 1 hour after surgery
  Measured in U/L
Blood urea nitrogen | 1 hour after surgery
  Measured in mg/dl
Creatinine | 1 hour after surgery
  Measured in mg/dl
Serum sodium level | 1 hour after surgery
  Measured in mmol/L
Serum potassium level | 1 hour after surgery
  Measured in mmol/L
Serum chloride | 1 hour after surgery
  Measured in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Jonghae Kim, M.D., Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea

REFERENCES:
- [Background] Alian AA, Galante NJ, Stachenfeld NS, Silverman DG, Shelley KH. Impact of lower body negative pressure induced hypovolemia on peripheral venous pressure waveform parameters in healthy volunteers. Physiol Meas. 2014 Jul;35(7):1509-20. doi: 10.1088/0967-3334/35/7/1509. Epub 2014 Jun 5. PMID 24901895
- [Background] Hocking KM, Sileshi B, Baudenbacher FJ, Boyer RB, Kohorst KL, Brophy CM, Eagle SS. Peripheral Venous Waveform Analysis for Detecting Hemorrhage and Iatrogenic Volume Overload in a Porcine Model. Shock. 2016 Oct;46(4):447-52. doi: 10.1097/SHK.0000000000000615. PMID 27070329
- [Background] Hocking KM, Alvis BD, Baudenbacher F, Boyer R, Brophy CM, Beer I, Eagle S. Peripheral i.v. analysis (PIVA) of venous waveforms for volume assessment in patients undergoing haemodialysis. Br J Anaesth. 2017 Dec 1;119(6):1135-1140. doi: 10.1093/bja/aex271. PMID 29028929
- [Background] Sileshi B, Hocking KM, Boyer RB, Baudenbacher FJ, Kohurst KL, Brophy CM, Eagle S. Peripheral venous waveform analysis for detecting early hemorrhage: a pilot study. Intensive Care Med. 2015 Jun;41(6):1147-8. doi: 10.1007/s00134-015-3787-0. Epub 2015 Apr 11. No abstract available. PMID 25862041